CLINICAL TRIAL: NCT02384759
Title: Phase II Randomized Trial Evaluting Aflibercept Associated With LV5FU2 Regimen as First Line Treatment of Non-resectalbe Metastatic Colorectal Cancers
Brief Title: Aflibercept +/- LV5FU2 in First Line of Non-resectalbe Metastatic Colorectal Cancers
Acronym: FOLFA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE25
Record Dates: First submitted 2015-01-28; First posted 2015-03-10 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Neoplasms
Keywords: cancer, colorectal,
MeSH Terms: conditions — Colorectal Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Aflibercept + LV5FU2
  Interventions: Drug: aflibercept; Drug: LV5FU2
- B (Active Comparator): LV5FU2
  Interventions: Drug: LV5FU2

INTERVENTIONS:
Drug: aflibercept
  Other Names: zaltrap
  Arms: A
Drug: LV5FU2

SUMMARY:
This is what the FFCD 11-01 - PRODIGE 25 trial proposes to study, as a preliminary for strategic studies evaluating the usefulness of including targeted therapeutics from the first line with aflibercept +/- LV5FU2.

DETAILED DESCRIPTION:
The aflibercept-5-FU combination has never been evaluated as yet. Aflibercept, at a dose of 4 mg/kg, has already been used in combination with 5-FU at the doses used in the simplified LV5FU2 regimen (folinic acid 400 mg/m2 IV in 90 min, then 5-FU 400 mg/m2 IV bolus on D1, followed by continuous perfusion of 5-FU 2,400 mg/m2 in 46h) (23) as part of the above-mentioned VELOUR trial, evaluating its combination with FOLFIRI (= simplified LV5FU2 + irinotecan). This trial was preceded by a phase I trial validating the doses used (24). It is therefore not necessary to perform a phase I trial if you use the same doses of 5-FU without irinotecan, within the context of a strategy for reducing toxicity in patients to be treated over a long period, and not search for the maximum tolerated dose of the combination.

The aflibercept-LV5FU2 combination can be useful for patients who will never be resectable or operable, and for whom 5-FU monotherapy can be suggested to delay the toxicities of combined chemotherapies. Within this context, it is possible for aflibercept to provide a survival benefit. The previous VELOUR trial (18) did not indicate that toxicity would have a major effect on quality of life and increase the hope of prolonged progression-free survival in the arm with aflibercept.

This is what the FFCD 11-01 - PRODIGE 25 trial proposes to study, as a preliminary for strategic studies evaluating the usefulness of including targeted therapeutics from the first line.

This trial will evaluate the efficacy of the combination and its tolerance by studying toxicities and quality of life. Quality of life will be studied via the EORTC questionnaire QLQ-C30.

The thymidylate synthase polymorphism type 2R2R-2R3R versus 3R3R seems to predict greater efficacy of 5-FU monotherapy. Stratification in this criterion will confirm or negate the prognostic or predictive nature of 5-FU efficacy linked to these polymorphisms.

The draft version of this trial has been studied and evaluated by the scientific council of the Fédération Francophone de Cancérologie Digestive (FFCD) then the Digestive Group of the Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC) within the framework of their Partnership for Research in Digestive Oncology (PRODIGE cooperation).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* General condition WHO ≤ 2
* Metastatic rectal or colonic adenocarcinoma, histologically proved on the primary tumour or a metastasis
* Metastases non-resectable and/or patient inoperable
* patients where a single agent chemotherapy combined with an anti-angiogenic agent is an appropriate approach
* At least one measurable target according to RECIST v1.1 criteria, no previously irradiated
* No previous treatment of the metastatic disease. Previous chemotherapy in an adjuvant situation completed 6 months or more before diagnosis of the metastasis is authorized.
* Adequate biological examination: Hb > or = 9 g/dl, polynuclear neutrophils > or = 1,500/mm3, platelets > or =100,000/mm3, total bilirubin < or = 1.5 x UNL, creatinine clearance, calculated according to Cockroft-Gault formula, > 50 ml/min creatininemia < 1.5 x UNL, ALP < 5 x UNL, transaminases < 5 x ULN, GGT< 5 x UNL
* Proteinuria (strip) < 2+; if > or = 2+, test proteinuria over 24 hours which must be ≤ 1 g.
* Central genotyping of thymidylate synthase (TS) in blood DNA
* Patients treated with anticoagulants (coumadin, warfarin) can be included if the INR can be closely monitored. A change in anticoagulant treatment for low molecular weight heparin is preferable in order to respect indications
* Signed written informed consent obtained prior to inclusion

Exclusion Criteria:

* Patients with a primary tumour in place and presenting clinical symptoms (occlusion, haemorrhage)
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* Uncontrolled hypercalcemia
* Uncontrolled hypertension (SBP > 150 mmHg and DBP > 100 mmHg) or history of hypertensive attacks or hypertensive encephalopathy
* Any progressive pathology not balanced over the past 6 months: hepatic insufficiency, renal insufficiency, respiratory insufficiency,
* Any of the following within 6 months prior to inclusion: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack.
* Any of the following within 3 months prior to inclusion: Grade 3-4 gastrointestinal bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event, wound or fractured bone
* Major surgery during the 28 days preceding the start of treatment
* Known acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease requiring antiretroviral treatment.
* Treatment with concomitant anticonvulsivant agents that are CYP3A4 inducers (phenytoin, phenobarbital, carbamazepine), unless discontinued >7 days.
* Anti-tumoral treatments other than the trial treatments (chemotherapy, targeted therapy, immunotherapy)
* Macronodular peritoneal carcinosis (risk of perforation)
* Known DPD deficit
* Prior history of malignant haemopathy or cancer except those treated more than 5 years ago and considered to be cured, in situ cervical carcinomas and treated skin cancers (excluding melanoma)
* Patients on new oral anticoagulant therapy (rivaroxaban XARELTOR, apixaban ELIQUIS, dagigatran PRADAXA except if relay by vitamine K antagonist therapy)
* Any contraindication to the treatments used in the trial
* Impossibility of undergoing medical monitoring during the trial for geographic, social or psychological reasons

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis LEGOUX, MD, Principal Investigator — ORLEANS - Centre Hospitalier La Source
Locations (58):
- France (58):
  - CH, Aix-en-Provence
  - CHU Amiens - Hôpital Nord, Amiens
  - Chu D'Angers, Angers
  - ICO, Angers
  - CH, Auxerre
  - CH de la Côte Basque, Bayonne
  - Centre D'Oncologie Et de Radiothérapie, Bayonne
  - CH, Béziers
  - Hôpital Avicenne, Bobigny
  - CHU APHP Hôpital Avicenne, Bobigny
  - CHU- Hôpital Saint André, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - CH - Hôpital Duchenne, Boulogne-sur-Mer
  - CH, Brive-la-Gaillarde
  - CHU Côte de Nacre, Caen
  - Ch, Chambéry
  - CH Public du Cotentin, Cherbourg
  - CHU Estaing, Clermont-Ferrand
  - CH Alpes Leman, Contamine-sur-Arve
  - Centre hospitalier Sud Francilien, Corbeil-Essonnes
  - Institut de cancérologie de Bourgogne - GRRECC, Dijon
  - CHU Le Bocage, Dijon
  - CH, Elbeuf
  - Chicas, Gap
  - CHD Vendée, La Roche-sur-Yon
  - CH Robert Boulin, Libourne
  - Clinique François Chénieux, Limoges
  - CHU, Limoges
  - Ch Longjumeau, Longjumeau
  - CH Hôpital du Surcoff, Lorient
  - Ch Saint Joseph - Saint Luc, Lyon
  - CHU APHM Hôpital Nord, Marseille
  - CHU APHM La Timone, Marseille
  - Hôpital Européen de Marseille, Marseille
  - CH, Meaux
  - CH, Montélimar
  - CHU - Hôtel Dieu, Nantes
  - Polyclinique de Languedoc, Narbonne
  - CHR La Source, Orléans
  - Saint-Louis CHU AP-HP Paris, Paris
  - CH, Perpignan
  - Hôpital Haut Leveque, Pessac
  - CHU Hôpital de la Milétrie, Poitiers
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Eugène Marquis, Rennes
  - CHU, Rouen
  - CARIO - Hôpital Privé des Côte d'Armor, Saint-Brieuc
  - ICO, Saint-Herblain
  - Polyclinique Côte Basque Sud, Saint-Jean-de-Luz
  - Ch Saintonges, Saintes
  - Centre de cancérologie Paris Nord, Sarcelles
  - CH de Bigorre, Tarbes
  - Hôpitaux du Leman, Thonon-les-Bains
  - CHU Hôpital Rangueil, Toulouse
  - Hôpital Trousseau, Tours
  - CHBA, Vannes
  - Institut Gustave Roussy, Villejuif
  - Hôpital Privé de Villeneuve d'Ascq, Villeneuve-d'Ascq

REFERENCES:
- [Result] Legoux JL, Faroux R, Barriere N, Le Malicot K, Tougeron D, Lorgis V, Guerin-Meyer V, Bourgeois V, Malka D, Aparicio T, Baconnier M, Lebrun-Ly V, Egreteau J, Khemissa Akouz F, Terme M, Lepage C, Boige V. First-Line LV5FU2 with or without Aflibercept in Patients with Non-Resectable Metastatic Colorectal Cancer: A Randomized Phase II Trial (PRODIGE 25-FFCD-FOLFA). Cancers (Basel). 2024 Apr 16;16(8):1515. doi: 10.3390/cancers16081515. PMID 38672597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2015 and September 2020, 117 patients were randomized in France
Groups:
- Aflibercept + LV5FU2: LV5FU2: LV5FU2 simplified every 2 weeks: folinic acid 400 mg/m2 IV over 90 min, then 5FU 400 mg/m2 IV bolus at D1, followed by continuous infusion of 5FU 2400 mg/m2 over 46 h.
  Aflibercept : Preceded or not by an IV infusion of aflibercept 4 mg/kg over 1 hour
- LV5FU2: LV5FU2 simplified every 2 weeks: folinic acid 400 mg/m2 IV over 90 min, then 5FU 400 mg/m2 IV bolus at D1, followed by continuous infusion of 5FU 2400 mg/m2 over 46 h.
Period: Overall Study
Arm/Group | Aflibercept + LV5FU2 | LV5FU2
Started | 59 | 58
Completed | 56 | 56
Not Completed | 3 | 2
Not completed — Patients not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline population is the mITT population meaning all the patients randomized into the study and having received at least one dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept + LV5FU2 | LV5FU2 | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 56 | 56 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.27 (5.43) | 80.23 (5.40) | 80.25 (5.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 35 | 33 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 56 | 56 | 112
Region of Enrollment [Number; unit: participants]
  France | 56 | 56 | 112

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective Was the Percentage of Patients Alive and Without Progression 6 Months After the Randomization.
Description: Progression was assessed by the investigator according to RECIST 1.1 criteria based on imaging studies performed every 8 weeks, even in case of deferred treatments. Clinical progressions, not confirmed on imaging, were not be counted in the primary endpoint
Time Frame: At 6 months after randomization
Population: Analysis population is the mITT population defined as all the patients randomized having received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept + LV5FU2 | LV5FU2
Number analyzed (Participants) | 56 | 56
Participants
  Percentage of patients alive without progression at 6 months | 30 | 30
  Percentage of patients with progression or death at 6 months | 26 | 26

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the patient's death (all causes). For alive patients, the date of the latest news was taken into account
Time Frame: Up to 3 years after the treatment start
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept + LV5FU2 | LV5FU2
Number analyzed (Participants) | 56 | 56
months | 21.85 [12.09 to 25.03] | 25.07 [19.84 to 31.93]

3. Secondary Outcome: Progression-free Survival (PPFS)
Description: It was defined as the time between t randomization and the date of the first radiological progression (RECIST 1.1 criteria) according to the investigator or death; Patients alive without progression were censored at the date of last news
Time Frame: up to 12 months after randomization
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept + LV5FU2 | LV5FU2
Number analyzed (Participants) | 56 | 56
months | 7.28 [5.59 to 8.25] | 7.23 [5.59 to 9.63]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment, on the average of 18 months. Death were monitored even the patient has stopped the study treatment (up to 3 years) whereas adverse events were monitored until the end of the study protocol (average of treatment=18 months)
Groups:
- LV5FU2: LV5FU2: LV5FU2 simplified every 2 weeks: folinic acid 400 mg/m2 IV over 90 min, then 5FU 400 mg/m2 IV bolus at D1, followed by continuous infusion of 5FU 2400 mg/m2 over 46 h.
Arm/Group | Aflibercept + LV5FU2 | LV5FU2
All-Cause Mortality (participants affected / at risk) | 37/56 | 36/56
Serious Adverse Events (participants affected / at risk) | 26/56 | 13/56
Other Adverse Events (participants affected / at risk) | 55/56 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + LV5FU2 (N=56) | LV5FU2 (N=56)
Thoracic Pain (Cardiac disorders) | 0 | 1
Auricular Fibrillation (Cardiac disorders) | 1 | 0
Cardiac insufficiency (Cardiac disorders) | 0 | 1
AVC (Nervous system disorders) | 2 | 0
Cephalgia (Nervous system disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Mental confusion (Psychiatric disorders) | 2 | 1
Veinous thromboembolic event (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 0
Haemorrhage (Blood and lymphatic system disorders) | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Fatigue (General disorders) | 6 | 0
Fever (General disorders) | 3 | 1
Burning (Injury, poisoning and procedural complications) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Cerebrovascular Ischemia (Nervous system disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + LV5FU2 (N=56) | LV5FU2 (N=56)
Anemia (Blood and lymphatic system disorders) | 37 | 42
Dorsalgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Hypertension (Vascular disorders) | 37 | 20
Anorexia (Metabolism and nutrition disorders) | 31 | 17
Fatigue (General disorders) | 49 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02384759/Prot_SAP_000.pdf